CLINICAL TRIAL: NCT06370767
Title: Enhancing Community Mobility in Individuals With Serious Mental Illnesses Through Peer-Facilitated Travel Training: A Two-armed Waitlist Controlled Trial
Brief Title: Peer Facilitated Waitlist Controlled Transportation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25634
Record Dates: First submitted 2024-03-27; First posted 2024-04-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Serious Mental Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either start the intervention program immediately, or be placed on an 8-week waitlist. Once randomized, the participant will again be randomized into a treatment condition: 1) peer-mediated bikeshare training intervention; or 2) peer-mediated public travel training intervention. 20 participants from each condition who have not opted out of being in the GPS subsample will be randomly assigned to be invited to a GPS subgroup.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bike-Share (Experimental): Participants in this arm will participate in an 8-week bikeshare training program, using Indego, the bike sharing service in Philadelphia. The first sessions will be aimed at increasing knowledge of the bike share program and the procedures for utilizing it successfully. Then participants will meet with a peer support specialist, who will help facilitate individualized route planning and independent ride support. Peer support specialists will use motivational interviewing during these individual sessions in order to help participants identify personally meaningful motivations for participation and to enhance their sense of self-efficacy.
  Interventions: Behavioral: Bike-Share Travel Training
- Public Transportation (Experimental): An established travel-training program developed for individuals with disabilities, including those with SMI, serves as the curriculum for the public transportation intervention arm. Participants will use SEPTA, the public transportation provider in Philadelphia and surrounding areas. We will offer an 8-week intervention which will include instruction on foundational skills needed to travel on public transportation and 1-on-1 direct training in using public transportation. Participants will meet twice weekly for direct instruction and role-playing sessions to cover the core components and the latter weeks of intervention will be focused on individual travel training instruction provided by the peer support interventionists, with participants and peer support interventionists meeting for two travel trips each week.
  Interventions: Behavioral: Public Transportation Travel Training
- Waitlist Control (No Intervention): Half of the participants in either arm (bike-share or public transportation) will be randomly assigned to either begin the intervention immediately, or be placed on a waitlist, serving as a control arm. The waitlist will be 8 weeks long, the same timeline as the intervention. After the eighth week, participants assigned to the waitlist will then begin the intervention for the next 8 weeks. Participants assigned to starting the intervention immediately will then be placed on the waitlist for the second-8 weeks of the total study enrollment.

INTERVENTIONS:
Behavioral: Bike-Share Travel Training — Half of the participants not assigned to the waitlist will begin the bike-share intervention arm immediately after the baseline research interview. The bike-share arm will last for 8 weeks and be delivered by a community peer specialist. Half of the participants assigned to the waitlist will begin the bike-share intervention arm after an 8-week waiting period.
  Arms: Bike-Share
Behavioral: Public Transportation Travel Training — Half of the participants not assigned to the waitlist or bike-share arm will begin the public transportation intervention arm immediately after the baseline research interview. The public transportation arm will last for 8 weeks and be delivered by a community peer specialist. Half of the participants assigned to the waitlist will begin the public transportation intervention arm after an 8-week waiting period.
  Arms: Public Transportation

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a peer-facilitated travel intervention in adults with serious mental illnesses. This project aims to address the following hypotheses:

1. Individuals with SMI receiving either of the two peer-mediated travel training transportation interventions will experience an increase in transportation self-efficacy and transportation skills.
2. Participants in the intervention arms will increase their transport utilization, participate in significantly more activities in the community, and make significantly more trips in the community.
3. Individuals with SMI receiving peer-mediated travel training interventions will retain post-test levels of community participation and self-efficacy 2 months after intervention.

Participants will be assigned to an 8-week travel-training intervention either using a bike-share program or public transportation. All participants will complete three data-collection research interviews.

DETAILED DESCRIPTION:
This project proposes using a two-armed, waitlist controlled trial to test the effectiveness of peer-facilitated travel interventions and their ability to enhance community mobility and increase feelings of self-efficacy in individuals with serious mental illness (SMI). The first intervention arm is an 8-week bikeshare intervention, which consists of individual trainings on using a bike sharing program; the second intervention arm is an 8-week public transportation intervention, which consists of individual trainings for using public transportation in the Philadelphia area. The investigators seek to enroll a total of 180 individuals from community mental health agencies in the Philadelphia area and expect recruitment to take 3 years. Eligible participants will be individuals who meet criteria indicating that they have an SMI, are between the ages of 18-65, and are both willing and able to learn to use public transportation and ride a bicycle. Data will be collected via face-to-face or web-based video call interviews at 3 time points: baseline, 2-months post-baseline, and 4-months post-baseline. Participants will also complete short surveys about their travel behaviors over the phone in the seven days after each interview. There will also be a subsample of participants who will provide additional GPS data.

ELIGIBILITY:
Inclusion Criteria:

* are between the ages of 18 and 65
* are diagnosed with a SMI (confirmed via the MINI)
* score at least an 8 on a travel skills assessment
* indicates that they can ride a bicycle
* have expressed interest in using a bikeshare and public transportation
* are able to provide informed consent

Exclusion Criteria:

* score less than 8 on a travel skills assessment
* express no interest in independent transportation
* are non-English speaking individuals
* are unable to provide consent
* are living in a setting where mobility and participation is restricted
* have a limiting physical condition that would prevent their ability to ride a bicycle independently

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Temple University Community Participation Measure | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  Measures engagement in 29 participation areas, if those areas are important to them, how often they did them and if it was enough, not enough, or too much. Higher reported frequency across a greater number of areas indicates higher rates of participation. Higher number of activities reported as being important and done enough indicate greater sufficiency of participation.
LASA Sedentary Behaviors Questionnaire | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This survey measures the time spent doing various activities that are usually completed while sitting down. For a 24-hour period on both weekdays and weekends, the reporting asks "How much time do you spend (from when you wake up until you go to bed) doing the following?" For this research, it will be used to measure changes in sedentary behaviors over time.
Transportation Appraisal Scale | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This measure assesses participants' ability to use public transportation and travel around their community. Items are asked on a 4-point scale, asking how much help is needed with various travel tasks, including reading schedules to plan a trip and knowing how to pay for transportation. For this research, it will be used to measure changes in transportation self-efficacy over time.
Indego Skills Survey | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This is an open-ended questionnaire to assess participants' skills with navigating the Indeo bike-sharing program in Philadelphia. Researchers give points to participants' responses on questions pertaining to the access, payment, and return of the bikes. For this research, it will be used to measure Indego skills at the time of the interview.
SEPTA Skills Survey | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  Similar to the Indego Skills Survey, this is an open-ended questionnaire to assess participants' skills with navigating Philadelphia's public transit system, SEPTA. Researchers give points to participants' responses on questions pertaining to the access, payment, and choosing the correct bus or subway stop. For this research, it will be used to measure SEPTA skills at the time of the interview
University of California, San Diego Performance-Based Skills Assessment (UPSA- Modified) | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This role-play measurement was designed for individuals with mental health challenges to assess participant's real-word abilities. The Transportation subscale uses a pitcutre of a bus schedule and asks the participant to correctly identify the departure, destination, and costs of rides. For this research, it will be used to measure SEPTA and bikeshare planning skills.
National Household Travel Survey | Administered daily for 7 days after baseline, 2-month, and 4-month follow-up interviews.
  This is a daily, self-report measure that captures the amount and types of trips a participant takes in one day. The log will be administered over the phone by a research assistant, asking how many trips were taken, the type of trip (medical appointment, work, social outing, etc), the mode of transportation (personal vehicle, public transit, bike, walk, etc) and the general location of the trip.
GPS | GPS data collection will last for 14 days after initial baseline interviews and another 14 days after completion of the 8-week intervention.
  A subsample of participants will carry a cellphone that will track their movements in the community using a GPS app. Outcome measures include: 1) number of unique destination, 2) total number of destinations, and 3) total distance traveled.
  A subsample of participants will carry a cellphone that will track their movements in the community using a GPS app. Outcome measures include: 1) number of unique destination, 2) total number of destinations, and 3) total distance traveled.
  A subsample of participants will carry a cellphone that will track their movements in the community using a GPS app. Outcome measures include: 1) number of unique destination, 2) total number of destinations, and 3) total distance traveled.
  A subsample of participants will carry a cellphone that will track their movements in the community using a GPS app. Outcome measures include: 1) number of unique destination, 2) total number of destinations, and 3) total distance traveled.

SECONDARY OUTCOMES:
Internalized Stigma of Mental Illness Inventory (ISMI) (Brief Version) | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This scale is designed to measure self-stigma among persons with psychiatric disorders. The brief measure takes the strongest items from each of the subscales of the full measure. The subscales and item examples include: Alienation (e.g. "Having a mental illness has spoiled my life"), Stereotype Endorsement (e.g., "Mentally ill people tend to be violent"), Discrimination Experience (e.g., "People discriminate against me because I have a mental illness"), Social Withdrawal (e.g., " I don't talk about myself as much because I don't want to burden others with my mental illness"), and Stigma Resistance (e.g., "I can have a good, fulfilling life, despite my mental illness") that is scored on a 4-point Likert scale. For this research, it will be used to measure changes in internalized stigma over time.
University of California, Los Angeles, Loneliness Scale | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  These 3 questions are only being given to people who report having a mental illness. The questions related to how often people feel socially isolated or lonely. Response options range from 1) hardly ever, 2) some of the time, and 3) often. Responses (3) indicate increased loneliness and more "hardly ever" responses indicate less loneliness.
Pearlin Mastery Scale (Coping) | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This is 7-item mastery scale to assess participants' feeling of control over their lives. Items are asked on a 4-point Likert scale and include statement like "I have little control over the things that happen to me" and "What happens to me in the future mostly depends on me." For this research, it will be used to measure changes in participants' abilities to cope with symptoms over time.
SF- 36 v2 | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This measure asks about health status and physical capability of daily activities. Participants are asked to rank their health over the last week, including experiences of pain, sickness, tiredness, and physical activities like walking or carrying. For this research, it will be used to measure self-perceived physical health.
The PERMA - Profiler Measure | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  The PERMA Profiler is based on the five pillars of wellbeing: positive emotion, engagement, relationships, meaning, accomplishment). Items are asked on a 10-pint scale and include items such as "How often do you schieve the important goals you have set for yourself?", "How lonely do you feel in your daily life?", and "To what extent do you feel loved?". For this research, it will be used to measure perceived quality of life.
Recovery Assessment Scale (RAS) | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  Three subscale from the RAS will be used: 1) reliance on others, 2) confidence and hope, and 3) willingness to ask for help. Responses range from strongly disagree (1) to strongly agree (5). Scores can range from 16-80 with higher scores indicating greater recovery, reliance on others, confidence, and willingness to ask for help.
Group Identification Scale (GIS) | Asked at baseline, 2-month, and 4-month follow-ups interviews.
  This scale measures intergroup relations and self-concept of group identification. Participants will be asked on a 7-point Likert scale how the agree or disagree with statements comparing them to other SEPTA and bikeshare riders. For this research, it will be used to measure participants' feeling of belonging in the groups of public transportation users, bikeshare, and their local community

CONTACTS AND LOCATIONS:
Locations (1):
- Pathways To Housing PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers, research institutions, or research databases for use in other studies. Per funder regulations, at the completion of the study all deidentified data will be transferred to ICPSR (https://www.icpsr.umich.edu/icpsrweb/) so that data can be used by others for additional analysis. Participants may request to have their data destroyed, but are notified at consent that de-identified data that has already been shared cannot be taken back or destroyed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study files will be kept for seven years after the last publication of the data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT06370767/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT06370767/ICF_001.pdf